CLINICAL TRIAL: NCT05773014
Title: Digital Versus Speculum Exams in Preterm Prelabor Rupture of Membranes: A Randomized Controlled Trial
Brief Title: Digital vs. Speculum Exams for PPROM
Acronym: MOCA
Status: Recruiting | Phase: Not Applicable | Type: Interventional
Sponsor: Washington University School of Medicine (Other)
Responsible Party: Sponsor
Allocation: Randomized | Model: Parallel | Masking: Single | Purpose: Other
Other Study IDs: 202301012
Record Dates: First submitted 2023-02-21; First posted 2023-03-17 (Actual); Last update posted 2026-01-05 (Actual); Status verified 2025-12

CONDITIONS: PPROM
Keywords: PPROM; speculum exam; preterm birth; preterm prelabor rupture of membranes
MeSH Terms: conditions — Preterm Premature Rupture of the Membranes; Premature Birth

STUDY DESIGN:
Who Masked: Outcomes Assessor
Oversight: Data Monitoring Committee: Yes | FDA-regulated Drug: No | FDA-regulated Device: No

ARMS (2):
- Speculum Exams (Active Comparator): If a patient requires cervical evaluation after PPROM, their cervix will be evaluated with a sterile speculum exam. A sterile speculum with lubricating jelly will be inserted into the patient's vagina to visualize the cervix and visually estimate cervical dilation and effacement.
  Interventions: Procedure: Speculum Exams
- Digital Exams (Active Comparator): If a patient requires cervical evaluation after PPROM, their cervix will be evaluated with a digital exam. The provider will wear sterile gloves with lubricating jelly and will palpate the cervix to assess cervical dilation, effacement, and station.
  Interventions: Procedure: Digital Exams

INTERVENTIONS:
Procedure: Speculum Exams — Same as arm
  Arms: Speculum Exams
Procedure: Digital Exams — Same as arm
  Arms: Digital Exams

SUMMARY:
After preterm prelabor rupture of membranes (PPROM)[breaking of the amniotic sac prior to 37 weeks gestation in pregnancy], patients are recommended for inpatient admission and close monitoring for complications including preterm labor, intraamniotic infection (infection of the sac around the baby), and placental abruption (separation of the placenta from wall of the uterus). When evaluation of cervical dilation is clinically indicated, obstetricians traditionally perform sterile speculum exams due to concern for decrease in pregnancy latency (length of time between breaking the water and delivery) with sterile digital exams in retrospective studies. These studies are concerning, however, by the indications for the exams and are at risk for confounding by indication. This is a randomized, non-inferiority trial to examine if sterile digital versus speculum exams effect latency of pregnancy in patients with PPROM.

ELIGIBILITY:
Inclusion Criteria:

* 22 weeks 0 days gestation to 33 weeks 5 days gestation
* Clinical or laboratory confirmation of PPROM
* At least 8 hours after rupture event
* English speaking

Notably, for patients <25 weeks, approach for enrollment will be deferred until after the patient has discussed their desires for fetal resuscitation with the care team and are at a gestational age where they would desire this resuscitation.

Exclusion Criteria:

* Contraindications to digital examination
* COVID-19 positive on admission

Sex: Female | Healthy Volunteers: Yes
Age Groups: Child, Adult, Older Adult
Gender Based: Yes — Patient must be pregnant
Enrollment: 86 (Estimated)
Dates: Start 2023-03-27 (Actual); Primary Completion 2027-03-01 (Estimated); Study Completion 2027-07-01 (Estimated)

PRIMARY OUTCOMES:
Pregnancy latency | up to 10 weeks
  time from admission to delivery

SECONDARY OUTCOMES:
Maternal chorioamnionitis | Prior to delivery
  Per criteria of American College of Obstetricians and Gynecologists (ACOG): includes fever greater than or equal to 100.4 degrees Farenheit plus an additional sign such as fundal tenderness, white blood cell count >15, purulent vaginal discharge, fetal tachycardia, or placental culture with finding of chorioamnionitis. Suspected chorioamnionitis can also be diagnosed with isolated fever >102.2 degrees Fahrenheit
Endomyometritis | Within 2 weeks of delivery
  Clinical diagnosis of uterine infection after delivery, typically with fever and fundal tenderness
Maternal sepsis | Within 2 weeks of delivery
  Defined as bacteremia with evidence of organ dysfunction
Maternal wound infections | Within 2 weeks of delivery
  As diagnosed by the clinicians
Maternal intensive care unit (ICU) admission | Within 2 weeks of delivery
  transfer to ICU or readmission to ICU
Maternal death | Within 2 weeks postpartum
  Death of mother
Composite neonatal morbidity | 28 days of life
  Need for respiratory support, neonatal sepsis, intraventricular hemorrhage, hypoxic ischemic encephalopathy, necrotizing enterocolitis, pneumonia, or neonatal demise
Length of neonatal intensive care unit (NICU) admission | Up to 1 year
  From delivery until discharge from the NICU
Need for respiratory support | 28 days of life
  One or more of the following: Continuous positive airway pressure (CPAP) or high-flow nasal cannula for at least 2 consecutive hours, supplemental oxygen with a fraction of inspired oxygen of at least 0.30 for at least 4 continuous hours, extracorporeal membrane oxygenation (ECMO), or mechanical ventilation
Neonatal sepsis at <72 hours of life | Within 72 hours of birth
  must be confirmed on blood culture
Neonatal sepsis at >72 hours of life | 28 days of life
  must be confirmed on blood culture
Neonatal intraventricular hemorrhage (IVH) | 28 days of life
  Seen on head ultrasound
Necrotizing enterocolitis (NEC) | 28 days of life
  As diagnosed by NICU team
Hypoxic ischemic encephalopathy | 28 days of life
  As diagnosed by NICU team
Neonatal pneumonia | 28 days of life
  As diagnosed by NICU team
Neonatal death | During NICU admission, up to 1 year
  As documented in the EMR
Patient satisfaction with exams | At delivery
  Survey regarding their experience with cervical exams

CONTACTS AND LOCATIONS:
Locations (1):
- Barnes Jewish Hospital, St Louis, Missouri, United States

IPD SHARING:
Plan to Share IPD: Undecided

REFERENCES:
- [Background] Sukcharoen N, Vasuratna A. Effects of digital cervical examinations on duration of latency period, maternal and neonatal outcome in preterm premature rupture of membranes. J Med Assoc Thai. 1993 Apr;76(4):203-9. PMID 8113640
- [Background] Alexander JM, Mercer BM, Miodovnik M, Thurnau GR, Goldenberg RL, Das AF, Meis PJ, Moawad AH, Iams JD, Vandorsten JP, Paul RH, Dombrowski MP, Roberts JM, McNellis D. The impact of digital cervical examination on expectantly managed preterm rupture of membranes. Am J Obstet Gynecol. 2000 Oct;183(4):1003-7. doi: 10.1067/mob.2000.106765. PMID 11035354
- [Background] Lewis DF, Major CA, Towers CV, Asrat T, Harding JA, Garite TJ. Effects of digital vaginal examinations on latency period in preterm premature rupture of membranes. Obstet Gynecol. 1992 Oct;80(4):630-4. PMID 1407885
- [Background] Singhal, S., Puri, M., & Gami, N. (2011). An analysis of factors affecting the duration of latency period and its impact on neonatal outcome in patients with PPROM. International Journal of Infertility and Fetal Medicine. 2012; 3(3): 87-91.